CLINICAL TRIAL: NCT02073461
Title: A Multicenter, Randomized, Double-blinded, Vehicle-controlled Parallel Group Efficacy and Safety Study of 2 Different Concentrations of CD1579 Gels Versus Vehicle in the Treatment of Acne Vulgaris.
Brief Title: Efficacy and Safety Study of 2 Different Concentrations of CD1579 Gels Versus Vehicle in the Treatment of Acne Vulgaris.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDT.07.SPR.27124
Record Dates: First submitted 2014-02-20; First posted 2014-02-27 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CD1579 2.5% (Experimental): Benzoyl Peroxide 2.5%
  Interventions: Drug: CD1579 2.5%
- CD1579 5% (Experimental): Benzoyl Peroxide 5%
  Interventions: Drug: CD1579 5%
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: CD1579 2.5%
  Other Names: Benzoyl Peroxide 2.5%
  Arms: CD1579 2.5%
Drug: CD1579 5%
  Other Names: Benzoyl Peroxide 5%
  Arms: CD1579 5%
Drug: Vehicle
  Arms: Vehicle

SUMMARY:
This study is to assess the efficacy and safety of two concentrations of CD1579 (2.5% and 5%) versus vehicle in the treatment of acne vulgaris in the Japanese patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at the age of 12 or older at the Screening visit.
* Those with clinical diagnosis of acne vulgaris with more than 20 noninflammatory lesions (open and closed comedones) and 12 to 100 (inclusive) inflammatory lesions (papules, pustules and nodules) on the face (forehead, both cheeks, nose and chin).

Exclusion Criteria:

* Those with more than two nodular acne lesions or any cysts.
* Those with the diagnosis of any acne conglobata, any acne fulminans, any chloracne, or any drug induced acne.
* Those who have clinically significant abnormal findings or conditions on skin other than acne such as atopic dermatitis, perioral dermatitis, or rosacea that potentially interfere with study assessments according to Investigator's judgment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Japan (6):
  - Galderma investigational site, Fukuoka, Fukuoka
  - Galderma investigational site, Amagasaki, Hyōgo
  - Galderma investigational site, Kobe, Hyōgo
  - Galderma investigational site, Nakano City, Tokyo
  - Galderma investigational site, Shibuya City, Tokyo
  - Galderma investigational site, Shinjuku, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- CD1579 2.5%: Benzoyl Peroxide 2.5%
  CD1579 2.5%
- CD1579 5%: Benzoyl Peroxide 5%
  CD1579 5%
Period: Overall Study
Arm/Group | CD1579 2.5% | CD1579 5% | Vehicle
Started | 79 | 78 | 79
Completed | 75 | 77 | 78
Not Completed | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CD1579 2.5% | CD1579 5% | Vehicle | Total
Number analyzed (Participants) | 79 | 78 | 79 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.1 (7.0) | 21.1 (5.6) | 21.0 (6.3) | 21.4 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 51 | 45 | 153
  Male | 22 | 27 | 34 | 83
Region of Enrollment [Number; unit: participants]
  Japan | 79 | 78 | 79 | 236

OUTCOME MEASURES:

1. Primary Outcome: Percent Changes From Baseline in Total Lesion Counts
Description: Median percent reductions from Baseline in total lesion count (ITT-LOCF)
Time Frame: Baseline - Week 12
Measure: Median (Full Range); unit: percent change
Arm/Group | CD1579 2.5% | CD1579 5% | Vehicle
Number analyzed (Participants) | 79 | 78 | 78
percent change | 58.3 [-243.7 to 100] | 65.9 [-41.0 to 100] | 25.5 [-180.7 to 88.9]

2. Secondary Outcome: Percent of Subjects With Adverse Events
Description: Adverse events which were observed in 5% or more patients with either group are listed.
Time Frame: up to 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | CD1579 2.5% | CD1579 5% | Vehicle
Number analyzed (Participants) | 79 | 78 | 79
percentage of participants
  % of subjects with AEs | 43.0 | 39.7 | 32.9
  Nasopharyngitis | 12.7 | 14.1 | 13.9
  Headache | 10.1 | 1.3 | 8.9
  Dysmenorrhea | 6.3 | 3.8 | 3.8

3. Secondary Outcome: Local Tolerability (Erythema)
Description: Highest severity of local tolerability scores worse than Baseline
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | CD1579 2.5% | CD1579 5% | Vehicle
Number analyzed (Participants) | 79 | 78 | 79
participants
  Mild | 12 | 18 | 5
  Moderate | 3 | 3 | 0
  Severe | 0 | 1 | 0

4. Secondary Outcome: Local Tolerability (Scaling)
Description: Highest severity of local tolerability scores worse than Baseline
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | CD1579 2.5% | CD1579 5% | Vehicle
Number analyzed (Participants) | 79 | 78 | 79
participants
  Mild | 15 | 25 | 8
  Moderate | 4 | 7 | 1

5. Secondary Outcome: Local Tolerability (Dryness)
Description: Highest severity of local tolerability scores worse than Baseline
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | CD1579 2.5% | CD1579 5% | Vehicle
Number analyzed (Participants) | 79 | 78 | 79
participants
  Mild | 20 | 33 | 10
  Moderate | 2 | 6 | 0

6. Secondary Outcome: Local Tolerability (Pruritus)
Description: Highest severity of local tolerability scores worse than Baseline
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | CD1579 2.5% | CD1579 5% | Vehicle
Number analyzed (Participants) | 79 | 78 | 79
participants
  Mild | 20 | 13 | 6
  Moderate | 6 | 7 | 1
  Severe | 1 | 2 | 0

7. Secondary Outcome: Local Tolerability (Stinging/Burning)
Description: Highest severity of local tolerability scores worse than Baseline
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | CD1579 2.5% | CD1579 5% | Vehicle
Number analyzed (Participants) | 79 | 78 | 79
participants
  Mild | 19 | 29 | 4
  Moderate | 6 | 7 | 1

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | CD1579 2.5% | CD1579 5% | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/78 | 1/79
Other Adverse Events (participants affected / at risk) | 34/79 | 31/78 | 26/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD1579 2.5% (N=79) | CD1579 5% (N=78) | Vehicle (N=79)
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD1579 2.5% (N=79) | CD1579 5% (N=78) | Vehicle (N=79)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema of eyelid (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) — General disorders and administration site conditions
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 2 (2) | 2 (2)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (11) | 11 (12) | 11 (12)
Oral herpes (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 8 (11) | 1 (7) | 7 (13)
Dysmenorrhoea (Reproductive system and breast disorders) | 5 (8) | 3 (4) | 3 (4)
Premenstrual syndrome (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No